CLINICAL TRIAL: NCT00961259
Title: Open-Label, Randomized, Single-Dose, 3-Arm, Crossover Pharmacokinetic and Bioequivalence Study of One 35 mg Fenofibric Acid Tablet and Three 35 mg Fenofibric Acid Tablets Versus One 105 mg Fenofibric Acid Tablet Under Fasting Conditions
Brief Title: Fasted Pharmacokinetic and Bioequivalency Study of Fenofibric Acid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-028-08-1017; R08-0057
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Results first posted 2009-11-05 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: healthy; pharmacokinetics; therapeutic equivalency; fenofibric acid
MeSH Terms: interventions — fenofibric acid; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fenofibric Acid 35 mg (1 x 35 mg tab) (Experimental): 1 x 35 mg tablet administered after an overnight fast of at least 10 hours
  Interventions: Drug: Fenofibric Acid 35 mg Tablet
- Fenofibric Acid 105 mg (3 x 35 mg tab) (Experimental): 3 x 35 mg tablets administered after an overnight fast of at least 10 hours
  Interventions: Drug: Fenofibric Acid 35 mg Tablet
- Fenofibric Acid 105 mg (1 x 105 mg tab) (Experimental): 1 x 105 mg tablet administered after an overnight fast of at least 10 hours
  Interventions: Drug: Fenofibric Acid 105 mg Tablet

INTERVENTIONS:
Drug: Fenofibric Acid 35 mg Tablet — 1 x 35 mg tablet administered after an overnight fast of at least 10 hours
  Arms: Fenofibric Acid 35 mg (1 x 35 mg tab)
Drug: Fenofibric Acid 35 mg Tablet — 3 x 35 mg tablets administered after an overnight fast of at least 10 hours
  Arms: Fenofibric Acid 105 mg (3 x 35 mg tab)
Drug: Fenofibric Acid 105 mg Tablet — 105 mg tablet administered after an overnight fast of at least 10 hours
  Arms: Fenofibric Acid 105 mg (1 x 105 mg tab)

SUMMARY:
This study will evaluate the pharmacokinetic linearity of a single 35 mg fenofibric acid dose and demonstrate the bioequivalence of three 35 mg fenofibric acid tablets (105 mg total single dose) to a single 105 mg fenofibric acid tablet in healthy adult volunteers when each dose is administered under fasted conditions. Safety and tolerability of these regimens will also be evaluated.

DETAILED DESCRIPTION:
This study will evaluate the pharmacokinetic linearity of a single 35 mg fenofibric acid dose and demonstrate the bioequivalence of three 35 mg fenofibric acid tablets (105 mg total single dose) to a single 105 mg fenofibric acid tablet in healthy adult volunteers when each dose is administered under fasted conditions. Fifty-four healthy, non-smoking, non-obese, 18-45 year old, male and female volunteers will be randomly assigned in a crossover fashion to receive each of three fenofibric acid dosing regimens in sequence with a 7 day washout period between dosing periods. On the morning of the first day of each dosing period, after an overnight fast of at least 10 hours, subjects will receive single doses of fenofibric acid (1 x 35 mg tablet), fenofibric acid (3 x 35 mg tablets - 105 mg total dose), or fenofibric acid (1 x 105 mg tablet). Fasting will continue for 4 hours after dose administration. Blood samples will be drawn from all participants prior to dosing and for 72 hours post-dose, at times sufficient to adequately define fenofibric acid pharmacokinetics. Subjects will be monitored throughout their participation for adverse reactions to the study drug and/or procedures. Seated blood pressure and pulse will be measured prior to each dose and approximately 2 hours after each dose to coincide with peak plasma concentrations. All adverse experiences, whether elicited by query, spontaneously reported, or observed by clinic staff, will be documented in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age
* Non-smoking
* Non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures)
* Body mass index (BMI) less than 30
* Medically healthy on the basis of medical history and physical examination
* Hemoglobin > or = to 12g/dL
* Completion of the screening process within 28 days prior to dosing
* Provision of voluntary written informed consent

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to fenofibric acid

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm.D., Principal Investigator — PRACS Institute

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-Four (54) non-obese, non-smoking, healthy adult volunteers from the community at large were enrolled.
Pre-assignment Details: One hundred and eight (108) subjects were screened. Thirty-six (36) subjects were screen failures. Of the remaining seventy-two (72) subjects, fifty-six (56) checked in and fifty-four (54) were enrolled.
Groups:
- Treatment Sequence ABC: On the morning of Day 1 after an overnight fast of at least 10 hours, each subject received one 35 mg fenofibric acid tablet (treatment A). After a 7 day washout period, on the morning of Day 8 after an overnight fast of at least 10 hours, each subject received three 35 mg fenofibric acid tablets (treatment B). After a 7 day washout period, on the morning of Day 15 after an overnight fast of at least 10 hours, each subject received one 105 mg fenofibric acid tablet (treatment C).
- Treatment Sequence BCA: On the morning of Day 1 after an overnight fast of at least 10 hours, each subject received three 35 mg fenofibric acid tablets (105 mg total dose, treatment B). After a 7 day washout period, on the morning of Day 8 after an overnight fast of at least 10 hours, each subject received one 105 mg fenofibric acid tablet (treatment C). After a 7 day washout period, on the morning of Day 15 after an overnight fast of at least 10 hours, each subject received one 35 mg fenofibric acid tablet (treatment A).
- Treatment Sequence CAB: On the morning of Day 1 after an overnight fast of at least 10 hours, each subject received one 105 mg fenofibric acid tablet (treatment C). After a 7 day washout period, on the morning of Day 8 after an overnight fast of at least 10 hours, each subject received one 35 mg fenofibric acid tablet (treatment A). After a 7 day washout period, on the morning of Day 15 after an overnight fast of at least 10 hours, each subject received three 35 mg fenofibric acid tablets (105 mg total dose, treatment B).
Period: First Intervention
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 18 | 18 | 18
Completed | 18 | 18 | 18
Not Completed | 0 | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 18 | 18 | 18
Completed | 18 | 17 (dropped due to concomitant medication used prior to admission.) | 18
Not Completed | 0 | 1 | 0
Not completed — due to concomitant medication used | 0 | 1 | 0
Period: Second Intervention
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 18 | 17 | 18
Completed | 18 | 17 | 18
Not Completed | 0 | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 18 | 17 | 18
Completed | 18 | 17 | 18
Not Completed | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 18 | 17 | 18
Completed | 18 | 17 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fenofibric Acid - Treatments A, B and C: All subjects received each of the three study regimens in a randomly assigned sequence of dosing periods. On the mornings of Days 1, 8 and 15 each subject received either one 35 mg fenofibric acid tablet (treatment A), three 35 mg fenofibric acid tablets (105 mg total dose, treatment B) or one 105 mg fenofibric acid tablet (treatment C).
Arm/Group | Fenofibric Acid - Treatments A, B and C
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.46 (7.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma. For the dosing group, Fenofibric Acid 35 mg (35 mg Dose-adjusted to 105 mg), the Cmax values were dose-adjusted in order to assess pharmacokinetic linearity.
Time Frame: serial pharmacokinetic blood samples drawn immediately prior to dosing and then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours after dose administration
Population: Pharmacokinetic analyses of fenofibric acid are based on 53 out of the 54 subjects who completed the study.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fenofibric Acid 35 mg (1 x 35 mg Tablet) - Treatment A; Fenofibric Acid 35 mg (35 mg Dose-adjusted to 105 mg): Each subject received one tablet of 35 mg fenofibric acid after an overnight fast of at least 10 hours.
- Fenofibric Acid 105 mg (3 x 35 mg Tablet) - Treatment B: Each subject received three tablets of 35 mg fenofibric acid after an overnight fast of at least 10 hours.
- Fenofibric Acid 105 mg (1 x 105 mg Tablet) - Treatment C: Each subject received one tablet of 105 mg fenofibric acid after an overnight fast of at least 10 hours.
Arm/Group | Fenofibric Acid 35 mg (1 x 35 mg Tablet) - Treatment A | Fenofibric Acid 35 mg (35 mg Dose-adjusted to 105 mg) | Fenofibric Acid 105 mg (3 x 35 mg Tablet) - Treatment B | Fenofibric Acid 105 mg (1 x 105 mg Tablet) - Treatment C
Number analyzed (Participants) | 53 | 53 | 53 | 53
ng/mL | 3,569.47 (685.12) | 10,708.40 (2,055.36) | 11,014.93 (2,033.94) | 11,202.87 (2,470.61)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule. For the dosing group, Fenofibric Acid 35 mg (35 mg Dose-adjusted to 105 mg), the [AUC(0-t)] values were dose-adjusted in order to assess pharmacokinetic linearity.
Time Frame: as for outcome 1
Population: Pharmacokinetic analyses of fenofibric acid are based on 53 out of the 54 subjects who completed the study.
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Fenofibric Acid 35 mg (1 x 35 mg Tablet) - Treatment A | Fenofibric Acid 35 mg (35 mg Dose-adjusted to 105 mg) | Fenofibric Acid 105 mg (3 x 35 mg Tablet) - Treatment B | Fenofibric Acid 105 mg (1 x 105 mg Tablet) - Treatment C
Number analyzed (Participants) | 53 | 53 | 53 | 53
ng-hr/mL | 49,419.89 (18,188.17) | 148,259.66 (54,564.52) | 131,976.95 (41,086.74) | 135,119.10 (42,326.25)

3. Primary Outcome: The Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity AUC(0-∞)
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant. For the dosing group, Fenofibric Acid 35 mg (35 mg Dose-adjusted to 105 mg), the AUC(0-∞) values were dose-adjusted in order to assess pharmacokinetic linearity.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours after drug administration.
Population: Pharmacokinetic analyses of fenofibric acid are based on 53 out of the 54 subjects who completed the study.
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Fenofibric Acid 35 mg (1 x 35 mg Tablet) - Treatment A | Fenofibric Acid 35 mg (35 mg Dose-adjusted to 105 mg) | Fenofibric Acid 105 mg (3 x 35 mg Tablet) - Treatment B | Fenofibric Acid 105 mg (1 x 105 mg Tablet) - Treatment C
Number analyzed (Participants) | 53 | 53 | 53 | 53
ng-hr/mL | 58,304.35 (20,877.56) | 174,913.04 (62,632.68) | 142,858.88 (45,554.44) | 147,555.58 (48,994.99)

ADVERSE EVENTS:
Description: 54 subjects were enrolled in this study. Several subjects dropped out of the study prior to receiving all interventions. 53 subjects were administered Fenofibric Acid (1 x 35mg tablets), 54 subjects were administered Fenofibric Acid 105 mg (3 x 35 mg Tablets), and 53 subjects were administered Fenofibric Acid 105 mg (1 x 105 mg Tablets).
Groups:
- Fenofibric Acid 35 mg (1 x 35 mg Tablet), Treatment A: Each subject received one tablet of 35 mg fenofibric acid after an overnight fast of at least 10 hours.
- Fenofibric Acid 105 mg (3 x 35 mg Tablet), Treatment B: Each subject received three (3) tablets of 35 mg fenofibric acid after an overnight fast of at least 10 hours.
- Fenofibric Acid 105 mg (1 x 105 mg Tablet), Treatment C: Each subject received one tablet of 105 mg fenofibric acid after an overnight fast of at least 10 hours.
Arm/Group | Fenofibric Acid 35 mg (1 x 35 mg Tablet), Treatment A | Fenofibric Acid 105 mg (3 x 35 mg Tablet), Treatment B | Fenofibric Acid 105 mg (1 x 105 mg Tablet), Treatment C
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/54 | 0/53
Other Adverse Events (participants affected / at risk) | 7/53 | 4/54 | 5/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibric Acid 35 mg (1 x 35 mg Tablet), Treatment A (N=53) | Fenofibric Acid 105 mg (3 x 35 mg Tablet), Treatment B (N=54) | Fenofibric Acid 105 mg (1 x 105 mg Tablet), Treatment C (N=53)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site hematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Orthodontic appliance complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days